CLINICAL TRIAL: NCT05234593
Title: Feasibility and Acceptability Study of a Powdered Multinutrient Formula in Children With Attention-Deficit/Hyperactivity Disorder and Emotional Dysregulation
Brief Title: Feasibility and Acceptability of Powdered Multinutrient Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jeanette Johnstone, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23379
Record Dates: First submitted 2022-01-19; First posted 2022-02-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lightning Stick (Other): Feasibility and acceptability
  Interventions: Dietary Supplement: EmpowerPlus Lightning Sticks

INTERVENTIONS:
Dietary Supplement: EmpowerPlus Lightning Sticks — multinutrient supplement containing vitamins, minerals, amino acids and antioxidants taken one Stick daily by dissolving the powder on or under the tongue

SUMMARY:
The study aims to test the feasibility and acceptability of 1) consumption of EMPowerplus Lightning Sticks, 2) at-home collection of blood and urine samples, and 3) remote visits and completion of online behavioral questionnaires.

DETAILED DESCRIPTION:
The study aims to test the feasibility and acceptability of 1) consumption of EMPowerplus Lightning Sticks, 2) at-home collection of blood and urine samples, and 3) remote visits and completion of online behavioral questionnaires. A limited number of blood samples will be used to generate cytokine data to test the ability to detect these molecules from the Tasso device-collected plasma. Parent and child questionnaire responses will examined for signals of change, but no formal statistical comparisons will be performed. This study will inform us whether a larger efficacy study is possible in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age inclusive of and between 7 and 16 years at the time of enrollment
2. Verbally willing to ingest one EmpowerPlus Lightning Stick daily
3. Attend all virtual study appointments and complete questionnaires
4. Have been previously enrolled in a multinutrient study OR complete a screening to match with participants from that study in terms of age and symptoms of ADHD and emotional dysregulation
5. Be medication and supplementation free (if supplement ingredient is contained in the Lightning Stick) prior to study initiation
6. Willing to collect blood and urine samples, once, at home.

Exclusion Criteria*:

1. Neurological disorder involving brain or other central function (e.g., history of, or suspected, intellectual disability, autism spectrum disorder, epilepsy, multiple sclerosis, narcolepsy) or other major psychiatric condition requiring hospitalization (e.g. significant mood disorder, active suicidal ideation, or psychosis), based on parent/guardian self-report of child's condition
2. Any serious medical condition, including inflammatory bowel disease, history of cancer, kidney or liver disease, hyperthyroidism, diabetes Type I or II
3. Known allergy to any ingredients of the intervention
4. Any known abnormality of mineral metabolism (e.g., Wilson's disease, hemochromatosis)
5. Taking any medication with primarily central nervous system activity, including stimulants used to treat symptoms of ADHD
6. Any disability that would interfere with participant answering questions verbally
7. Non-English speaking
8. Pregnancy or sexually active at baseline. *Exclusion criteria will be based on parent/guardian report on child. If the parent/guardian reports medical exclusion criteria, or concerns about eligibility, data provided by parent/guardian will be confirmed by review of medical records with release of information signed by parent/guardian. Potential participants may be reviewed virtually by study physician in the case of any concerns about participation.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by count of remaining Sticks | week 6
  Feasibility will be determined if consumption of one Lightning Stick daily is achieved when greater than or equal to 80% of provided Sticks were taken.
  Measured by count of remaining (unused) Sticks.
Abbreviated Acceptability Rating Profile - 7 questions on a 6-point Likert scale | week 6
  Acceptability of taking the Lightning Sticks will be measure through 7 questions with a 6-point Likert-scale, (range: Strongly Disagree to Strongly Agree) Acceptability will be achieved if greater than or equal to 70% of children and parents report that taking powdered multinutrients is acceptable, at or above the Agree range.

SECONDARY OUTCOMES:
Feasibility measured by count of participants who provide blood using the Tasso device | once, at baseline
  At-home collection of blood with the Tasso device will be considered feasible if greater than or equal to 70% of children provide the sample.
Acceptability measured by a 'yes' response to their preference of using the Tasso device instead of a lab-based blood draw | once, at baseline
  Acceptability will be measured if greater than or equal to 70% of children and parents state they preferred the Tasso at-home collection method instead of going to a lab to provide the blood sample.
Feasibility measured by count of participants who provide the dried urine sample | once, at baseline
  At-home collection of dried urine samples will be considered feasible if greater than or equal to 70% of children provide the sample.
Acceptability measured by a 'yes' response to their preference of using the at-home dried urine sample collection method instead of a lab-based urine sample collection method | once, at baseline
  Acceptability will be measured if greater than or equal to 70% of children and parents state they preferred the at-home dried urine collection method instead of going to a lab to provide the urine sample.
Feasibility of remote study visits measured by count of participants who complete all online remote study visits | week 6
  Feasibility will be determined if greater than or equal to 70% of parents/guardians complete all three remote visits
Acceptability measured by a 'yes' response to their preference of completing online remote study visits instead of in-person study visits | week 6
  Acceptability will be measured if greater than or equal to 70% of parents state they preferred completing online remote study visits instead of in-person study visits
Monitor participants for side effects by count of 'yes' if listed symptoms are new or have increased in severity, using the question format from the Pediatric Adverse Events Rating Scale | week 6
  Parent and child report of side effects, including: headache, dry mouth, sleep disruptions, nausea, irritability, fatigue, anxiety, changes in appetite, skin rash, migraines, and other (specify what symptom).

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Johnstone, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No